CLINICAL TRIAL: NCT05058235
Title: Comparison Of Effects Of Active Release Technique And Bent Leg Raise On Hamstring Flexibility In Patients With Knee Osteoarthritis
Brief Title: Comparison of Active Release Technique and Bent Leg Raise In Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00853 Syeda Nayab Sheeraz
Record Dates: First submitted 2021-08-23; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
Keywords: Active Release Technique; Bent leg raise; Hamstring flexibility
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique (Experimental): Hot pack, TENS, Quadriceps Isometric strengthening, Active Release Technique
  Interventions: Other: Active Release Technique
- Bent leg raise (Active Comparator): Hot pack, TENS, Quadriceps Isometric strengthening, Bent leg raise
  Interventions: Other: Bent leg raise

INTERVENTIONS:
Other: Active Release Technique — Moist Hot pack 10 mins/1 set/ (6 days/ week), TENS 20 mins/1 set/ (6 days/ week), Quadriceps Isometric Strengthening 5 sec hold, 10 reps/ 1 set/(6 days/ week), Active release Technique 5 reps/ 1 set/ (6 days/ week)
  A total of 2 weeks (12 sessions, 6 sessions/ week) were given each consisting of 40 mins.
  Arms: Active Release Technique
Other: Bent leg raise — Moist Hot pack 10 mins/1 set/ (6 days/ week), TENS 20 mins/1 set/ (6 days/ week), Quadriceps Isometric Strengthening 5 sec hold, 10 reps/ 1 set/(6 days/ week), Bent leg raise 5 sec hold/ 5 sec stretch/ 3 reps/ 1 min rest interval/ 1 set/ (6 days/ week).
  A total of 2 weeks (12 sessions, 6 sessions/ week) were given each consisting of 40 mins.
  Arms: Bent leg raise

SUMMARY:
The objective of the study was to compare the effects of active release technique and bent leg raise on hamstring flexibility, functional outcomes, and pain in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee Osteoarthritis is a common progressive degenerative joint disease. Muscular weakness and other structural abnormalities can cause low back pain. Hamstring muscle being a postural muscle has an increased tendency to become tight. In this study, participants with knee osteoarthritis having hamstring tightness were included. Active Release Technique and Bent Leg Raise technique have been used to increase flexibility in hamstrings in these patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of Knee Osteoarthritis
* Hamstring length less than 160 degrees
* Minimum history of 3 months
* Willing to participate

Exclusion Criteria:

* Patients who have passive knee extension more than 160 degrees
* Patients with less than 3 months history
* Patients who have osteoarthritis of other than the knee joint
* Patients with history of fracture
* Patients with post surgical history

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Hamstring flexibility | 12 days
  Changes from baseline, Hamstring flexibility was measured through passive knee extension test with the help of Goniometer. Normal value of knee extension angle is 180 degrees. Values decreased than 160 degree represents hamstring tightness.

SECONDARY OUTCOMES:
Functional outcome | 12 days
  Changes from baseline, Functional outcome was taken through western Ontario McMaster Universities Osteoarthritis Index tool. It comprises three sections containing 24 items. Score ranges from 0 to 96. 0 representing a healthy state and higher scores indicating worst health.
Pain on Visual analogue Scale | 12 days
  Changes from baseline, Pain was measured through Visual Analogue Scale. It comprises of a continuous scale of 10cm line. 0 to 4mm represents "no pain", 5mm to 44mm indicates "mild pain", whereas 45mm to 74mm indicates "moderate pain" and continues to the range of "worst pain" between 75mm to 100 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, Phd, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Noor Physio and Sports Injury Clinic, G-8 Markaz, Islamabad, Federal
  - Riphah Rehabilitation Center, Westridge campus, Potohar Tower, Peshawar Road, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No